CLINICAL TRIAL: NCT02915627
Title: Study to Examine the Hemodynamic Responses in Hemodialysis Patients to Blood Flow Restriction Using Non-pneumatic Anti-shock Garments
Brief Title: Hemodynamic Responses in Hemodialysis Patients to Blood Flow Restriction Using Non-pneumatic Anti-shock Garments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Chris McIntyre, Professor of Medicine, UWO, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 108183
Record Dates: First submitted 2016-09-14; First posted 2016-09-27 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Blood Pressure
Keywords: Antishock Garment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy participants (Active Comparator): Non chronic kidney disease (CKD) participants. Intervention: Application of antishock garment. Participants will be examined for two 15 minute intervals with and without the anti-shock garments applied. During each 15 minute interval, echocardiograms will be performed.
  Interventions: Device: Application of Antishock garment
- CKD patients not on dialysis (Active Comparator): CKD 4/5 patients not on Dialysis- Intervention: Application of antishock garment. Participants will be examined for two 15 minute intervals with and without the anti-shock garments applied. During each 15 minute interval, echocardiograms will be performed.
  Interventions: Device: Application of Antishock garment
- CKD patients on Dialysis (Active Comparator): Patients having haemodialysis treatment at least 3 times per week at a London Health Sciences Centre facility-Intervention: Application of antishock garment. Participants will be examined for two 15 minute intervals with and without the anti-shock garments applied. During each 15 minute interval, echocardiograms will be performed.
  Interventions: Device: Application of Antishock garment

INTERVENTIONS:
Device: Application of Antishock garment — anti-shock garments are applied. Participants will then be examined for two 15 minute intervals with and without the anti-shock garments applied. During each 15 minute interval, echocardiograms will be performed.

SUMMARY:
Study comparing different groups of people and how they respond to application of the non-pneumatic anti-shock garments. Investigators will divide all recruited participants into three groups based on health status (group 1: hemodialysis patients; group 2: patients with severe chronic kidney disease but not on dialysis; group 3: healthy participants with no clinically known kidney disease). Each group, which will comprise of 10 people, will receive the same treatment using the non-pneumatic anti-shock garments.

DETAILED DESCRIPTION:
Primary Aim: To determine how blood flow restriction to the lower extremities using non-pneumatic anti-shock garments affects hemodynamic and cardiovascular parameters such as blood pressure in Hemodialysis (HD) patients while they are not on dialysis.

Investigators propose a pilot study to assess the effects of blood flow restriction using non-pneumatic anti-shock garments in HD patients while they are not on dialysis.

Outcomes: The primary objective will be a measurement of blood pressure upon application of the non-pneumatic anti-shock garments.

Secondary outcomes will include the following: baroreflex sensitivity; trends in beat-to-beat blood pressure upon application of the anti-shock garments; patient tolerability of the non-pneumatic anti-shock garments, ejection fraction via echocardiogram analyses.

ELIGIBILITY:
Inclusion Criteria:

Healthy participants

1. Male and female, age≥18 years old
2. No clinical diagnosis of CKD

CKD patients not on dialysis

1. Male and female, age≥18 years old
2. Stage 4 or Stage 5 CKD patients

CKD patients on dialysis

1. Male and female, age≥18 years old
2. Patients having haemodialysis treatment at least 3 times per week at a London Health Sciences Centre facility

Exclusion Criteria:

1. Not meeting inclusion criteria
2. Severe heart failure (New York Heart Association grade IV)
3. Pulmonary hypertension
4. Mitral stenosis
5. Cardiac transplant recipients
6. Mental incapacity to consent
7. Declined to participate
8. Absence of lower limbs or lower limb injury
9. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-11; Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Assessment of blood pressure changes with and without garment application | Participants will be examined for two 15 minute intervals with and without the anti-shock garments applied. During each 15 minute interval, echocardiograms will be performed.
  a measurement of blood pressure upon application of the non-pneumatic anti-shock garments

SECONDARY OUTCOMES:
Assessment of changes in Baroreflex Sensitivity with and without garment application. | Participants will be examined for two 15 minute intervals with and without the anti-shock garments applied. During each 15 minute interval, echocardiograms will be performed.
  baroreflex sensitivity; upon application of the anti-shock garments;
Assessment of changes in trends in beat to beat blood pressure with and without garment application. | Participants will be examined for two 15 minute intervals with and without the anti-shock garments applied. During each 15 minute interval, echocardiograms will be performed.
  trends in beat-to-beat blood pressure upon application of the anti-shock garments
Assessment of participant tolerability with garment application. | Participants will be examined for a 15 minute interval with the anti-shock garments applied. During each 15 minute interval, echocardiograms will be performed.
  Participant tolerability of the anti-shock garments
Assessment of changes in ejection fraction with and without garment application. | Participants will be examined for two 15 minute intervals with and without the anti-shock garments applied. During each 15 minute interval, echocardiograms will be performed.
  changes in ejection fraction upon application of anti-shock garment

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marinovich R, Li Z, Tamasi T, Quinn K, Wong S, McIntyre CW. Hemodynamic response to non-pneumatic anti-shock compression garments in patients with renal dysfunction. BMC Nephrol. 2020 Jan 14;21(1):15. doi: 10.1186/s12882-019-1680-8. PMID 31937266